CLINICAL TRIAL: NCT06445036
Title: Tunisian Clinical Registry on Hypoparathyroidism and Pseudo-hypoparathyroidism
Acronym: THYPARS
Status: Not yet recruiting | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Société Tunisienne D'endocrinologie De Diabétologie Et Des Maladies Métaboliques (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-015-THYPARS
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hypoparathyroidism; Pseudo Hypoparathyroidism
Keywords: Hypoparathyroidism; Pseudo Hypoparathyroidism; Clinical Registry; Endocrinology; Parathyroid gland
MeSH Terms: conditions — Hypoparathyroidism; Pseudohypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational, multicenter, national, cross-sectional study aiming to describe the epidemiological clinical, biological and therapeutic profile of patients suffering from defect in secretion (hypoparathyroidism) or action (pseudo-hypoparathyroidism) of parathyroid hormone.

DETAILED DESCRIPTION:
Endocrinologists from both sectors (public and private) are participating in the study. Data will be captured electronically by DACIMA Clinical Suite, according to FDA 21 CFR part 11 (Food and Drug Administration 21 Code of Federal Regulations part 11), HIPAA (Health Insurance Portability and Accountability Act) & ICH (International Conference on Harmonisation) requirements.

ELIGIBILITY:
Inclusion Criteria:

* Hypoparathyroidism defined by low serum calcium < 2.2 mmol/l (< 88 mg/l) associated with inadequate PTH (low or normal) and normal creatinine

Exclusion Criteria:

* Cervical surgery < 6 months.
* Transient (neonatal, etc.) or functional (dysmagnesemia, etc.) hypoparathyroidism.
* Other causes of hypocalcemia: vitamin D deficiency, chronic renal failure, etc.
* Familial hypocalcemia hypercalciuria.
* Pseudo-pseudo-hypoparathyroidism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients suffering from hypoparathyroidism and/or pseudo hypoparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-27 (Estimated); Primary Completion 2025-07-27 (Estimated); Study Completion 2025-07-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary hypoparathyroidism | Day 1
  Number of subjects with primary hypoparathyroidism at enrollment
Incidence of congenital hypoparathyroidism | Day 1
  Number of subjects with congenital hypoparathyroidism at enrollment
Incidence of acquired hypoparathyroidism | Day 1
  Number of subjects with acquired hypoparathyroidism at enrollment
Incidence of secondary hypoparathyroidism | Day 1
  Number of subjects with secondary hypoparathyroidism at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Nabila Rekik Mejdoub, MD, Study Chair — Société Tunisienne D'endocrinologie De Diabétologie Et Des Maladies Métaboliques
Locations (1):
- Société Tunisienne D'endocrinologie De Diabétologie Et Des Maladies Métaboliques, Sfax, Tunisia, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of Société Tunisienne D'endocrinologie De Diabétologie Et Des Maladies Métaboliques — https://endocrino-tunisie.com/